CLINICAL TRIAL: NCT06315725
Title: A Randomized Cross-Over Study to Investigate the Effect of the Non-Nutritive Sweetener Sucralose on Glucose Metabolism in Patients with Type 1 Diabetes
Brief Title: Effect of Artificial Sweetener (AFS) on Glucose Metabolism in Patients with Type 1 Diabetes (T1D)
Acronym: AFS_T1D
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dana Small, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2024-10504
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes (T1D); Healthy Subjects
Keywords: Type 1 Diabetes; Artificial Pancreas; Artificial Sweeteners; Non-Nutritive Sweeteners; Cross-Over; Taste Perception; Indirect Calorimetry; Insulin; Glucose Metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Sweet taste perception with/without sweet taste blockade — In our study, we will use our four different novel flavored beverages, with and without a sweet taste blockade.

SUMMARY:
The goal of this randomized crossover study is to test the prediction that consuming carbohydrates will affect insulin release differently depending on whether Non-Nutritive Sweeteners (NNSs) are consumed simultaneously. We aim to determine whether the predicted effects are associated with oral or post-oral sweet taste receptor signaling,. Our study will focus on patients diagnosed with type 1 diabetes (T1D) who are using an artificial pancreas (AP) system, as it allows us to monitor glucose and insulin levels over time.

Participants will drink four different flavored beverages, some with sweet taste blockade and some without, in a counter-balanced order. They will then rate the sweetness of each beverage, and we will collect data from their AP system to monitor insulin and glucose level.

To achieve this, we will conduct a pilot study to assess the effectiveness and best timing of sweet taste blockade in healthy individuals. Insights gained from the pilot study will inform the main study.

Sucralose will be used as the NNS, maltodextrin as the carbohydrate, and Gymnema Sylvestre (GS) as the sweet taste receptor blocker.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of T1D
* HbA1C ≤ 8 %
* Insulin pump therapy
* Adults of any gender or biological sex aged 18-45 years old,
* Body Mass Index (BMI) between 18.5-29.9 kg/m,
* Non-smokers,
* English or French speaker. ●. Who can consume chicken and fish

Exclusion Criteria:

* A major medical diagnosis that could potentially influence metabolic dysfunction
* A major medical diagnosis other than T1D,
* Alcohol or substance use disorder,
* Eating disorder or history of malabsorptive syndrome,
* Inflammatory bowel disease,
* Self-reported impairment in taste or smell,
* A known taste or smell dysfunction (e.g., anosmia),
* Active pregnancy and/or lactation,
* Food allergies or intolerances,
* Dislike of the test beverages,
* History of bariatric surgery at any point in the past ●. Regular consumer of Gymnema sylvestre

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: For the pilot study, 10 healthy participants will be recruited. For the main study, 15 potential participants with T1D will be recruited.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness and optimal time course of sweet test blockade on sweet taste perception in healthy individuals | from enrollment to the end of treatment at 4 weeks
  our aim is to test whether the impact of consuming NNS with carbohydrates on glucose metabolism is related to oral or post-oral sweet taste receptor signaling.
Mean plasma glucose, basal and bolus insulin changes in individuals with T1D on AP following beverage consumption. | From enrollment to the end of treatment at 4 weeks
  Consuming NNS alongside carbohydrates affects glucose metabolism differently compared to carbohydrates alone in participants with type 1 diabetes (T1D) using an artificial pancreas (AP) system for exogenous insulin production

SECONDARY OUTCOMES:
Resting Energy Expenditure (REE) and nutrient partitioning changes in individuals with T1D on AP following beverage consumptionT1D on AP following beverage consumption | from enrollment to the end of treatment at 4 weeks
  To test whether the co-ingestion of the NNS with carbohydrate can result in changes in post-ingestion metabolism, we plan to employ indirect calorimetry (IC) to evaluate resting energy expenditure (REE) before and after flavoured beverages consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Innovative Medicine, The Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada